CLINICAL TRIAL: NCT00923676
Title: Effect of Fenofibrate and Rosuvastatin on Sexual Dysfunction in Hyperlipidemic Patients. A Randomized Trial
Brief Title: Treatment of Hyperlipidemia and Sexual Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Dario Giugliano, Prof of Endocrinology, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DGMM/03/2007
Record Dates: First submitted 2009-06-15; First posted 2009-06-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Sexual Dysfunction; Hyperlipidemia
Keywords: Hyperlipidemia; LDL-cholesterol; HDL-cholesterol; triglycerides; IIEF; FSFI; Male and female sexual dysfunctions
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Hyperlipidemias | interventions — Fenofibrate; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fenofibrate (Active Comparator): Fenofibrate pills
  Interventions: Drug: fenofibrate
- Rosuvastatin (Active Comparator): Rosuvastatin pills
  Interventions: Drug: Rosuvastatin
- fenofibrate + rosuvastatin (Active Comparator): fenofibrate pills + rosuvastatin pills
  Interventions: Drug: fenofibrate + rosuvastatin

INTERVENTIONS:
Drug: fenofibrate — pill 145 mg, 145 mg/day, for 12 months
  Arms: Fenofibrate
Drug: Rosuvastatin — pills of 10 mg, 10 mg/day, 12 months
  Arms: Rosuvastatin
Drug: fenofibrate + rosuvastatin — fenofibrate 145 mg/day + rosuvastatin 10 mg/day for 12 months
  Arms: fenofibrate + rosuvastatin

SUMMARY:
Hyperlipidemias are frequently associated with and are considered an important cause of erectile dysfunction in men. This association has been attributed to the impairment of blood flow through endothelium-dependent relaxation in smooth muscle cells of corpus cavernosum. Basic science and human research suggest that the vascular pathophysiology of male and female sexual dysfunction may be similar, as the first phase of the female sexual response is mediated by a combination of vasocongestive and neuro-muscular event which include increased clitoral length and diameter, as well as increased vaginal lubrication, wall engorgement and luminal diameter. The investigators have shown that women with hyperlipidemia had a higher prevalence of sexual dysfunction as compared with age-matched women without hyperlipidemia.

The aim of this study was to asses the effect of anti-hyperlipidemic drugs (fenofibrate and rosuvastatin, single or in combination) on validated indices of sexual function in hyperlipidemic men and women with sexual dysfunction at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Low-density lipoprotein (LDL)-cholesterol levels > 160 mg/dL, high-density lipoprotein (HDL)-cholesterol levels < 50 mg/dL (for women) and < 40 mg/dl (for men), or triglyceride levels > 150 mg/dL.
* Stable heterosexual partner relationship for the preceding 6 months.

Exclusion Criteria:

* Pregnancy or less than 8 weeks postpartum.
* Diabetes mellitus (fasting glucose > 126 mg/dl.
* Uremia.
* Multiple sclerosis.
* Chronic alcoholism (intake of ≥ 500g/wk).
* Cancer.
* Psychiatric problems.
* Symptomatic cardiovascular disease.
* Gynecological surgery.
* Pelvic trauma.
* Polycystic ovarian syndrome.
* Abnormal thyroid function.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2008-04; Primary Completion 2015-10 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
International index of erectile dysfunction (IIEF) in men and Female sexual function index (FSFI) in women | Baseline, 6 months, 12 months

SECONDARY OUTCOMES:
Blood lipids, inflammatory markers | Baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD,PhD, Principal Investigator — Department of Geriatrics and Metabolic Diseases, Second University of Naples, Italy
Locations (1):
- Department of Geriatrics and Metabolic Diseases, Naples, Italy

REFERENCES:
- [Background] Esposito K, Ciotola M, Maiorino MI, Giugliano F, Autorino R, De Sio M, Cozzolino D, Saccomanno F, Giugliano D. Hyperlipidemia and sexual function in premenopausal women. J Sex Med. 2009 Jun;6(6):1696-1703. doi: 10.1111/j.1743-6109.2009.01284.x. Epub 2009 Apr 23. PMID 19453904